CLINICAL TRIAL: NCT01766960
Title: Altered Drug Disposition and Biomarkers for Diagnosis of Chronic Inflammatory Liver Disease.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of North Carolina, Greensboro (Other)
Responsible Party: Principal Investigator, Sidney Barritt, MD, Assistant Professor of Medicine, University of North Carolina, Chapel Hill
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-1599; 550KR41202 (Other Grant/Funding Number: NC TraCS Institute)
Record Dates: First submitted 2013-01-04; First posted 2013-01-11 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Fatty Liver
Keywords: Bile acids; Pharmacokinetics
MeSH Terms: conditions — Fatty Liver | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy volunteers (Experimental): Subjects will be asked to fast overnight. Upon presentation, FibroScan procedure with CAP will be conducted and baseline and postprandial bile acid profile will be assessed. Then, intravenous morphine will be administered and the pharmacokinetic profile will be assessed over 8 hours.
  Interventions: Other: High fat meal; Drug: Morphine
- Advanced nonalcoholic fatty liver disease patients (Experimental): Subjects will be asked to fast overnight. Upon presentation, FibroScan procedure with CAP will be conducted and baseline and postprandial bile acid profile will be assessed. Then, intravenous morphine will be administered and the pharmacokinetic profile will be assessed over 8 hours.
  Interventions: Other: High fat meal; Drug: Morphine

INTERVENTIONS:
Other: High fat meal — A high fat breakfast will be administered to induce gall bladder emptying.
Drug: Morphine — Five milligrams of intravenous morphine will be administered.

SUMMARY:
One-third of the U.S. population suffers from non-alcoholic fatty liver disease (NAFLD). NAFLD is caused by diabetes and obesity, and is becoming more common. Although many people have this disease, the change in how the liver handles drugs and compounds in the body has not been studied. The purpose of this study is to investigate how advanced NAFLD changes the ability of the liver to handle both endogenous and exogenous compounds.

ELIGIBILITY:
Inclusion Criteria:

General:

* Man or woman between 18 and 65 years of age
* Negative pregnancy test for women of childbearing potential
* Negative urine drug screen

Healthy Subjects:

* Normal liver function tests
* Normal kidney function and lipid panel

Nonalcoholic Steatohepatitis Patients:

* Recent liver biopsy with nonalcoholic fatty liver disease activity score at least 4

Exclusion Criteria:

General:

* History of significant alcohol use (>20 g/day) and/or illicit drug use
* Inability to abstain from alcohol for 48 prior to study
* Use of drugs associated with a clinical or histological picture consistent with fatty liver disease or NASH for more than 12 consecutive weeks in the year prior to screening; these include amiodarone, tamoxifen, methotrexate, glucocorticoids, anabolic steroids, tetracyclines, estrogens (at doses greater than those used for hormone replacement) or valproate/valproic acid
* Type 2 diabetes treated with oral agents other than metformin; these include secretagogues, thiazolidinediones, alpha-glucosidase inhibitors, exenatide and pramlintide.
* Current or recent use of bile acid sequestrants, bile acid derivatives (i.e. ursodiol) or fibric acid derivatives.
* Current use of antioxidants such as silymarin, vitamin C, glutathione, or non-prescribed complementary alternative medications (including dietary supplements, megadose vitamins, herbal preparations, and special teas) within 30 days prior to screening.
* Previous liver biopsy that demonstrated presence of cirrhosis.
* Radiologic imaging consistent with cirrhosis or portal hypertension.
* Serum creatinine of 2.0 mg/dL or greater, or on dialysis, at screening.
* History of immunologically mediated disease (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, severe psoriasis, rheumatoid arthritis) that could affect the assessment of biomarkers (bile acids or inflammation).
* History of bariatric surgery.
* BMI > 45 kg/m^2 at screening.
* Any known hypersensitivity to opiates, opiate antagonists, or ondansetron.

Healthy Subjects:

* Taking concomitant medications, both prescription and non-prescription (including herbal products and over-the-counter medications), other than oral contraceptives and multivitamins (women stabilized on hormonal methods of birth control will be allowed to participate)
* History or other evidence of liver disease in the opinion of the study investigators.
* BMI > 30 kg/m^2 at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-11; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of morphine and its hepatically derived metabolites. | 8 hours post dose
  Morphine will be administered as a 5-min IV infusion. Pharmacokinetic profiles of morphine and morphine metabolites will be quantified in the serum over the 8-hour sampling period. Non-compartmental analysis will be performed using Pharsight Phoenix software, comparing the following parameters between healthy subjects and patients with advanced NAFLD. The maximal concentration, time of maximal concentration, elimination half-life, area under the curve, and systemic and renal clearances will be calculated for both morphine and the glucuronide metabolites. Volume of distribution and metabolic clearance will be calculated for morphine.

SECONDARY OUTCOMES:
Bile acid profile | Pre- and postprandially
  The bile acid profile in healthy and diseased subjects will be assessed following an 8 hour fast and every 30 min for 2 hours following a high fat breakfast. At each of the 5 time points, serum concentrations of total and selected individual bile acid species will be quantified and compared between healthy subjects and patients with advanced NAFLD. Comparison of the bile acid profile, comprised of all selected bile acids, between subjects and patients will pose as the primary endpoint for this outcome.
FibroScan with Controlled Attenuation Parameter (CAP) Software | No preparation (fasting) required-consumption of large meals prior to the Fibroscan procedure is not advised
  FibroScan is more sensitive method to identify less severe scarring of liver tissue when compared to liver ultrasound and contrary to liver biopsy, it is not invasive. In this study, Fibroscan will be used to assess the extent of liver fibrosis in both healthy volunteers and patients diagnosed with NAFLD and the CAP software will be used to estimate fat liver content. These findings will be correlated with changes in morphine disposition and bile acid profile observed in the study participants as described above.

CONTACTS AND LOCATIONS:
Overall Officials: Alfred S Barritt, MD, Principal Investigator — University of North Carolina, Chapel Hill; Kim LR Brouwer, PharmD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- North Carolina Clinical and Translational Research Center, Chapel Hill, North Carolina, United States